CLINICAL TRIAL: NCT04773938
Title: Endoscopic Third Ventriculostomy for Adults With Hydrocephalus: Creating a Prognostic Model for Success - A Retrospective Multicenter Study
Brief Title: Endoscopic Third Ventriculostomy for Adults: A Prognostic Model for Success
Acronym: NordicETV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sondre Tefre, MD, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: NordicETV
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Hydrocephalus
Keywords: Endoscopic third ventriculostomy; Adult
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic Third Ventriculostomy for Adults with Hydrocephalus: Creating a Prognostic Model for Success - A Retrospective Multicenter Study

Background: Endoscopic third ventriculostomy (ETV) is becoming an increasingly widespread treatment for hydrocephalus, but most of the research is based on paediatric populations. The ETV Success Score (ETVSS) was developed in 2009 to predict the outcome of ETV in children. There is no similar tool for predicting outcome in adults.

Objective: The purpose of this study is to create a prognostic model to predict the success of ETV for adult patients with hydrocephalus

Methods: The study will adhere to the TRIPOD reporting guidelines and will be conducted as a retrospective chart review of all patients ≥18 years old treated with ETV at the participating centres between Jan 1st, 2010 and Dec 31st, 2018. Data collection is conducted locally in REDCap. Univariate analyses will be used to identify several strong predictors to be included in a multivariate logistic regression model. The model will be validated using K-fold cross validation. Discrimination will be assesses using AUROC and calibration with calibration belt plots.

Expected outcomes: The ability to predict who will benefit from an ETV will allow better primary patient selection both for ETV and shunting. This would reduce additional second procedures due to primary treatment failure. A success score specific for adults could also be used as a communication tool to provide better information and guidance to patients.

DETAILED DESCRIPTION:
Endoscopic Third Ventriculostomy for Adults with Hydrocephalus: Creating a Prognostic Model for Success - a retrospective multicenter study

Background:

The most common treatment for hydrocephalus is a ventriculoperitoneal shunt (VPS), to divert excess CSF from the ventricles to be absorbed in the peritoneum. The treatment can be applied to different aetiologies of hydrocephalus, but there is a high complication risk both short and long term. A retrospective review of 17,035 adult patients who had undergone their first VPS surgery for hydrocephalus, report that one third (33.4%) of the patients experienced at least one complication, during the follow up (3.9 years), and 22% required revision. 21.4% of the complications occurred within the first year. Another revew of 683 adult patients, found that 32% experienced shunt failure, with 74% occurring within 6 months.

Endoscopic third ventriculostomy (ETV) is an alternative treatment option, creating a passage between the ventricles and the subarachnoid space, by perforating the floor of the third ventricle. It is minimally invasive and leaves no mechanical foreign body behind, thereby avoiding many of the implant complications associated with VPS.

The overwhelming majority of research on endoscopic third ventriculostomy (ETV) is conducted in paediatric or mixed paediatric/adult populations. ETV Success Score (ETVSS) was created in 2009 to predict the outcome of ETV treatment in children. The ETVSS consists of three factors: age, aetiology and shunt history. Based on these factors a score from 0-90 is given, representing the predicted probability of successful ETV outcome 6 months postoperatively. The ETVSS was tested in a mixed population of 168 patients with a mean age of 40 years (range 3-85 years) and found to have inadequate discrimination with an AUC of 0.61 but good calibration.

The ETVSS is based on paediatric populations, and the age differentiation stops after the patient has reached 10 years. 50 out of a possible 90 points are given if the patient is more than 10 years old, making this parameter in the ETVSS redundant when used in adults. Furthermore, the ETVSS does not include several common aetiologies for adult hydrocephalus such as idiopathic normal pressure hydrocephalus (iNPH), subarachnoid haemorrhage (SAH) and long-standing overt ventriculomegaly in adults (LOVA). Previous shunt treatment seems to play an important role in adults as well. A review of 163 adult patients reported an overall success rate of 80%, with patients treated with ETV as the primary treatment faring significantly better than those with a previous shunt, at 87% and 65% respectively.

Radiological findings are not included in the ETVSS, and although most radiological signs of obstruction are subjective evaluations based on the observer's experience, some quantifiable signs have been identified. Downward bowing of the third ventricular floor has been identified as a strong predictor of ETV success. The bowing was measured by placing a line through the chiasma to the top of the mesencephalon or the mamillary bodies. Downward bowing was defined as inferior displacement of the third ventricle floor below this line.

Although there are a few studies analysing long-term ETV survival in adults, most are in paediatric or mixed populations. The existing long-term series on adult patients show most failures occurring shortly after the procedure although late failures are reported. Kaplan Meier curves for ETV survival have an initial steep decline, followed by a gradual fall-off before it seems to stabilise with few failures after a certain point. By determining the composition of patient characteristics these three different parts of the curve. The initial fall off is hypothesised to represent patients without benefit of the procedure and significant symptoms requiring early re-operation. The second group are also ineffective from the beginning, but present with more chronic symptomatology giving more time to evaluate the effect before re-operation. The failures occurring in the stable part of the curve represents initial success with a late closure of the stoma.

With ETV becoming an increasingly widespread treatment for adult hydrocephalus there is a need for a new prognostic model specific for this patient population. The ability to predict who will benefit from an ETV will allow better primary patient selection both for ETV and shunting, reduce additional second procedures because of primary treatment failure, and possibly prevent further unnecessary procedures.

Objective

The purpose of this study is to create a prognostic model to predict the short-term success of ETV for adult patients with hydrocephalus.

Speciﬁc aims for this research project is to:

1. Identify factors associated with both success and failure of ETV in adults, to establish a prognostic model.
2. Report on ETV success rates, complications and survival in adult patients at the partici-pating centres.

A success score specific for adults will improve patient selection and can also be used as a communication tool to provide better information and guidance to patients. The prognostic model will be tested in a future prospective study conducted at the participating centres. As well as follow up on the study population in the future to report long-term outcomes.

Hypotheses

Main hypothesis:

An adult ETVSS can be created based on patient demographics, symptomatology, aetiology, shunt history and radiologic ﬁndings.

Secondary hypotheses:

* Age is still a relevant factor but has the inverse effect in adults with less successful out-comes with older age.
* Aetiology and shunt history have prognostic value but must be recalibrated to reﬂect the spectrum of hydrocephalus conditions in adults.
* It is possible to develop a radiological hydrocephalus classiﬁcation and scoring system providing additional prognostic value.
* There are different characteristics in the failures occurring during the different phases seen on the Kaplan Meier survival curve.

Methodology

Study design:

The study will be conducted as a retrospective review of electronic patient charts and will adhere to the TRIPOD guidelines in the development of the prediction model. A multivariate logistic regression model will be used to identify prognostic factors for success of ETV treatment. This model is expected to be simplified to include only 3 to 4 strong predictors to make it useful in daily clinical practice.

Data collection and monitoring:

Each of the participating centres will be responsible for the data collection in a standardised database, that will include demographic information (date of birth, sex) and details on aetiology (haemorrhage, infection, tumour or cyst, trauma, congenital or idiopathic), symptomatology (acute and chronic symptoms), previous shunt treatment (number revisions, cause of malfunction, duration of shunt treatment), radiological investigations (visible obstruc-tion or radiological signs of obstruction), surgical details (date, equipment, technique, concur-rent procedures, following procedures) complications (intra- and postoperative, length of stay) and follow-up (at 3-12 months and most recent) All ETVs performed at the participating centres will be entered in the database and then includ-ed or excluded based on the below delineated criteria. Reason for exclusion will be registered, and the in-built tools in REDCap used to uncover missing data.

Oversight:

Approval from the Danish Patient Safety Authority (Styrelsen for Patientsikkerhed) and The Danish Data Protection Agency (Datatilsynet) has been granted.

Definition of ETV-success Success is defined as clinical improvement at first follow up, with no further CSF-diversion procedures within the first year of follow up. Clinical improvement will be registered based on the records from the first available follow up, but also include patients where the ETV was deemed ineffective before the patient was discharged or where a second procedure was per-formed during the same admission. If the patient's chart leaves any doubt when registering if the patient's symptoms improved postoperatively, it should be registered as "not improved". If the patient receives further CSF-diversion procedures during the first year, the ETV is considered a failure. Implantation of ICP-monitoring equipment does not render the ETV unsuccessful, un-less it is followed by CSF-diversion. Patients undergoing repeat ETV are counted as failures when calculating the success rate, but results are registered in order to determine the efficacy of re-ETVs. Additional CSF-diversion procedures will be registered for the entire observation pe-riod (beyond the first year) to determine long-term ETV-survival.

Sample size:

There is no clear consensus on the required sample size for prognostic models based on retrospective data. However, the paediatric ETVSS was based on 618 paediatric patients, using 70% (455) of the population for the creation of the model and the remaining 30% (163) for validation. Based on this the minimum number of patients required, is approximately 500. There is no upper limit, as more patients would give a better foundation for the prediction model, especially in the rarer patient categories such as iNPH or hydrocephalus caused by infection or SAH. approximately 220 adult ETV patients have been identified in Copenhagen 2010-2018. With cooperation between several centres the sample should easily meet the minimum required sample size and provide the necessary power to create a robust prognostic model. Approximately 250 ETVs are expected from each of the participating countries, resulting in 1000 patients. The model will be tested in a separate prospective study.

Statistical Analysis:

Patient demographics, aetiology and shunt history, as well as complications, will be summarised using descriptive statistics. The patient's symptoms are categorised as 'improved' or 'not improved' following treatment. If the patient requires subsequent CSF diversion procedures or fails to show clinical improvement, the ETV is considered a failure. Each of the proposed predictors are analysed in a univariate statistical analysis and are subsequently included in a multivariate logistic regression model to construct a uniﬁed prediction model. Statistical signiﬁcance is deﬁned at p<0.05. The model will be validated using K-fold cross validation. Discriminative ability will be assessed using AUROC and calibration using calibration belt plots. Significant missing data will be handled using multiple imputation. Time to ETV failure will be analysed using Kaplan-Meier curves.

Financial plan:

As this is a retrospective chart review, limited funds are required. ST has been partially funded by the Lundbeck Foundation and the Hjerne- og Nervekirurgisk Forskningspulje, Rigshospitalet. No other specific funding has been received for this study.

ELIGIBILITY:
Inclusion Criteria:

* ETV procedure performed
* ≥18 years old at time of first ETV

Exclusion Criteria:

* <18 years old at time of first ETV
* Permanent intraventricular foreign bodies left behind after the ETV. eg. Shunt or stents. Temporary external ventricular drains, ICP-monitoring probes or ligated shunts where the ventricular drain is removed, are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all first time ETV performed at the participating centres between January 1st 2010 and December 31st 2018.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
ETV success | Evaluated 1 year after operation
  The procedure is considered successful if the patient experience clinical improvement at first follow up and receives no further CSF diversion procedures, within one year of the initial procedure.

SECONDARY OUTCOMES:
ETV survival | From procedure to latest documented follow-up, adressed up to 31 dec. 2020.
  Time to ETV failure, using Kaplan-Meier analysis is calculated based on date of another CSF diversion procedure or the time a lack of clinical improvement is registered, whichever may come first.
ETV related adverse events | Up to 3 months after operation.
  Descriptive statistics of all registered intraoperative and postoperative complications, deficits and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Sondre Tefre, Principal Investigator — Department of Neurosurgery, Copenhagen University Hospital Rigshospitalet; Marianne Juhler, Study Director — Department of Neurosurgery, Copenhagen University Hospital Rigshospitalet
Locations (19):
- Denmark (4):
  - Department of Neurosurgery, Aalborg University Hospital, Aalborg
  - Department of Neurosurgery, Aarhus University Hospital, Aarhus
  - Department of Neurosurgery, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Department of Neurosurgery, Odense University Hospital, Odense
- Finland (4):
  - Department of Neurosurgery, Helsinki University Hospital and University of Helsinki, Helsinki
  - Department of Neurosurgery NeuroCenter Kuopio University Hospital, Kuopio
  - Department of Neurosurgery, Oulu University Hospital, Oulu, Finland & Research Unit of Clinical Neuroscience, Oulu University, Oulu
  - Neurocenter, Department of Neurosurgery and Turku Brain Injury Center, Turku University Hospital and University of Turku, Turku
- Norway (5):
  - Department of Neurosurgery, Haukeland University Hospital, Bergen
  - Department of Neurosurgery, Oslo University Hospital Rikshospitalet, Oslo
  - Department of Neurosurgery, Oslo University Hospital Ullevål, Oslo
  - Department of Neurosurgery, University Hospital of North Norway, Tromsø
  - Department of Neurosurgery, St. Olavs University Hospital, Trondheim
- Sweden (6):
  - Department of Neurosurgery, Sahlgrenska University Hospital, Gothenburg
  - Department of Neurosurgery in Linköping, and Department of Biomedical and Clinical Sciences, Linköping University, Linköping
  - Department of Neurosurgery, Lund University Hospital, Lund
  - Department of Neurosurgery, Karolinska University Hospital, Stockholm
  - Department of Neurosurgery, Umeå University Hospital, Umeå
  - Department of Neurosurgery, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
The study is conducted as part of the Nordic Young Neurosurgeons Research Collaborative (NYNReC). Data is available upon reasonable request. Interested parties must apply in writing through nynrec.org including plan for analysis and dissemination of findings. Application will be evaluated by the NYNReC Committee and study lead. A request for access may be declined if the proposal lacks clarity or a satisfactory methodology.
URL: https://www.nynrec.org/

REFERENCES:
- [Background] Kulkarni AV, Drake JM, Mallucci CL, Sgouros S, Roth J, Constantini S; Canadian Pediatric Neurosurgery Study Group. Endoscopic third ventriculostomy in the treatment of childhood hydrocephalus. J Pediatr. 2009 Aug;155(2):254-9.e1. doi: 10.1016/j.jpeds.2009.02.048. Epub 2009 May 15. PMID 19446842
- [Background] Reddy GK, Bollam P, Caldito G, Willis B, Guthikonda B, Nanda A. Ventriculoperitoneal shunt complications in hydrocephalus patients with intracranial tumors: an analysis of relevant risk factors. J Neurooncol. 2011 Jun;103(2):333-42. doi: 10.1007/s11060-010-0393-4. Epub 2010 Sep 15. PMID 20842407
- [Background] Merkler AE, Ch'ang J, Parker WE, Murthy SB, Kamel H. The Rate of Complications after Ventriculoperitoneal Shunt Surgery. World Neurosurg. 2017 Feb;98:654-658. doi: 10.1016/j.wneu.2016.10.136. Epub 2016 Nov 5. PMID 27826086
- [Background] Reddy GK, Bollam P, Shi R, Guthikonda B, Nanda A. Management of adult hydrocephalus with ventriculoperitoneal shunts: long-term single-institution experience. Neurosurgery. 2011 Oct;69(4):774-80; discussion 780-1. doi: 10.1227/NEU.0b013e31821ffa9e. PMID 21508873
- [Background] Grand W, Leonardo J, Chamczuk AJ, Korus AJ. Endoscopic Third Ventriculostomy in 250 Adults With Hydrocephalus: Patient Selection, Outcomes, and Complications. Neurosurgery. 2016 Jan;78(1):109-19. doi: 10.1227/NEU.0000000000000994. PMID 26295500
- [Background] Bouras T, Sgouros S. Complications of endoscopic third ventriculostomy. J Neurosurg Pediatr. 2011 Jun;7(6):643-9. doi: 10.3171/2011.4.PEDS10503. PMID 21631203
- [Background] Dusick JR, McArthur DL, Bergsneider M. Success and complication rates of endoscopic third ventriculostomy for adult hydrocephalus: a series of 108 patients. Surg Neurol. 2008 Jan;69(1):5-15. doi: 10.1016/j.surneu.2007.08.024. PMID 18054606
- [Background] Labidi M, Lavoie P, Lapointe G, Obaid S, Weil AG, Bojanowski MW, Turmel A. Predicting success of endoscopic third ventriculostomy: validation of the ETV Success Score in a mixed population of adult and pediatric patients. J Neurosurg. 2015 Dec;123(6):1447-55. doi: 10.3171/2014.12.JNS141240. Epub 2015 Jul 24. PMID 26207604
- [Background] Foley RW, Ndoro S, Crimmins D, Caird J. Is the endoscopic third ventriculostomy success score an appropriate tool to inform clinical decision-making? Br J Neurosurg. 2017 Jun;31(3):314-319. doi: 10.1080/02688697.2016.1229744. Epub 2016 Sep 14. PMID 27624099
- [Background] Breimer GE, Sival DA, Brusse-Keizer MG, Hoving EW. An external validation of the ETVSS for both short-term and long-term predictive adequacy in 104 pediatric patients. Childs Nerv Syst. 2013 Aug;29(8):1305-11. doi: 10.1007/s00381-013-2122-8. Epub 2013 May 5. PMID 23644629
- [Background] Durnford AJ, Kirkham FJ, Mathad N, Sparrow OC. Endoscopic third ventriculostomy in the treatment of childhood hydrocephalus: validation of a success score that predicts long-term outcome. J Neurosurg Pediatr. 2011 Nov;8(5):489-93. doi: 10.3171/2011.8.PEDS1166. PMID 22044375
- [Background] Waqar M, Ellenbogen JR, Stovell MG, Al-Mahfoudh R, Mallucci C, Jenkinson MD. Long-Term Outcomes of Endoscopic Third Ventriculostomy in Adults. World Neurosurg. 2016 Oct;94:386-393. doi: 10.1016/j.wneu.2016.07.028. Epub 2016 Jul 17. PMID 27436208
- [Background] Dlouhy BJ, Capuano AW, Madhavan K, Torner JC, Greenlee JD. Preoperative third ventricular bowing as a predictor of endoscopic third ventriculostomy success. J Neurosurg Pediatr. 2012 Feb;9(2):182-90. doi: 10.3171/2011.11.PEDS11495. PMID 22295925
- [Background] Kehler U, Regelsberger J, Gliemroth J, Westphal M. Outcome prediction of third ventriculostomy: a proposed hydrocephalus grading system. Minim Invasive Neurosurg. 2006 Aug;49(4):238-43. doi: 10.1055/s-2006-950382. PMID 17041837
- [Background] Isaacs AM, Bezchlibnyk YB, Yong H, Koshy D, Urbaneja G, Hader WJ, Hamilton MG. Endoscopic third ventriculostomy for treatment of adult hydrocephalus: long-term follow-up of 163 patients. Neurosurg Focus. 2016 Sep;41(3):E3. doi: 10.3171/2016.6.FOCUS16193. PMID 27581315
- [Background] Hong S, Hirokawa D, Usami K, Ogiwara H. The long-term outcomes of endoscopic third ventriculostomy in pediatric hydrocephalus, with an emphasis on future intellectual development and shunt dependency. J Neurosurg Pediatr. 2019 Jan 1;23(1):104-108. doi: 10.3171/2018.7.PEDS18220. Epub 2018 Oct 12. PMID 30497212
- [Background] Dewan MC, Lim J, Shannon CN, Wellons JC 3rd. The durability of endoscopic third ventriculostomy and ventriculoperitoneal shunts in children with hydrocephalus following posterior fossa tumor resection: a systematic review and time-to-failure analysis. J Neurosurg Pediatr. 2017 May;19(5):578-584. doi: 10.3171/2017.1.PEDS16536. Epub 2017 Mar 10. PMID 28291428
- [Background] Stovell MG, Zakaria R, Ellenbogen JR, Gallagher MJ, Jenkinson MD, Hayhurst C, Mallucci CL. Long-term follow-up of endoscopic third ventriculostomy performed in the pediatric population. J Neurosurg Pediatr. 2016 Jun;17(6):734-8. doi: 10.3171/2015.11.PEDS15212. Epub 2016 Feb 12. PMID 26870897
- [Background] Faggin R, Calderone M, Denaro L, Meneghini L, d'Avella D. Long-term operative failure of endoscopic third ventriculostomy in pediatric patients: the role of cine phase-contrast MR imaging. Neurosurg Focus. 2011 Apr;30(4):E1. doi: 10.3171/2011.1.FOCUS10303. PMID 21456920
- [Background] Beuriat PA, Puget S, Cinalli G, Blauwblomme T, Beccaria K, Zerah M, Sainte-Rose C. Hydrocephalus treatment in children: long-term outcome in 975 consecutive patients. J Neurosurg Pediatr. 2017 Jul;20(1):10-18. doi: 10.3171/2017.2.PEDS16491. Epub 2017 Apr 21. PMID 28430083
- [Background] Sacko O, Boetto S, Lauwers-Cances V, Dupuy M, Roux FE. Endoscopic third ventriculostomy: outcome analysis in 368 procedures. J Neurosurg Pediatr. 2010 Jan;5(1):68-74. doi: 10.3171/2009.8.PEDS08108. PMID 20043738
- [Background] Kadrian D, van Gelder J, Florida D, Jones R, Vonau M, Teo C, Stening W, Kwok B. Long-term reliability of endoscopic third ventriculostomy. Neurosurgery. 2005 Jun;56(6):1271-8; discussion 1278. doi: 10.1227/01.neu.0000159712.48093.ad. PMID 15918943
- [Background] Gangemi M, Mascari C, Maiuri F, Godano U, Donati P, Longatti PL. Long-term outcome of endoscopic third ventriculostomy in obstructive hydrocephalus. Minim Invasive Neurosurg. 2007 Oct;50(5):265-9. doi: 10.1055/s-2007-990305. PMID 18058641
- [Background] Vulcu S, Eickele L, Cinalli G, Wagner W, Oertel J. Long-term results of endoscopic third ventriculostomy: an outcome analysis. J Neurosurg. 2015 Dec;123(6):1456-62. doi: 10.3171/2014.11.JNS14414. Epub 2015 Jul 31. PMID 26230473
- [Background] Vogel TW, Bahuleyan B, Robinson S, Cohen AR. The role of endoscopic third ventriculostomy in the treatment of hydrocephalus. J Neurosurg Pediatr. 2013 Jul;12(1):54-61. doi: 10.3171/2013.4.PEDS12481. Epub 2013 May 17. PMID 23682819
- [Background] Rahme R, Rahme RJ, Hourani R, Moussa R, Nohra G, Okais N, Samaha E, Rizk T. Endoscopic third ventriculostomy: the Lebanese experience. Pediatr Neurosurg. 2009;45(5):361-7. doi: 10.1159/000257525. Epub 2009 Nov 11. PMID 19907200
- [Background] Gliemroth J, Kasbeck E, Kehler U. Ventriculocisternostomy versus ventriculoperitoneal shunt in the treatment of hydrocephalus: a retrospective, long-term observational study. Clin Neurol Neurosurg. 2014 Jul;122:92-6. doi: 10.1016/j.clineuro.2014.03.022. Epub 2014 Mar 26. PMID 24908225
- [Background] Woodworth GF, See A, Bettegowda C, Batra S, Jallo GI, Rigamonti D. Predictors of surgery-free outcome in adult endoscopic third ventriculostomy. World Neurosurg. 2012 Sep-Oct;78(3-4):312-7. doi: 10.1016/j.wneu.2011.09.018. Epub 2011 Nov 7. PMID 22120264
- [Derived] Tefre S, Lilja-Cyron A, Arvidsson L, Bartek J, Corell A, Forsse A, Glud AN, Hamdeh SA, Hansen FL, Huotarinen A, Johansson C, Kamarainen OP, Korhonen T, Kotkansalo A, Mansoor NM, Mendoza Mireles EE, Miscov R, Munthe S, Nittby-Redebrandt H, Obad N, Pedersen LK, Posti J, Raj R, Satopaa J, Stahl N, Tetri S, Tobieson L, Juhler M. Endoscopic third ventriculostomy for adults with hydrocephalus: creating a prognostic model for success: protocol for a retrospective multicentre study (Nordic ETV). BMJ Open. 2022 Jan 31;12(1):e055570. doi: 10.1136/bmjopen-2021-055570. PMID 35105647